CLINICAL TRIAL: NCT02317341
Title: Effect of Ketamine on Fatigue Following Cancer Therapy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 150037; 15-NR-0037
Record Dates: First submitted 2014-12-13; First posted 2014-12-16 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03-18

CONDITIONS: Cancer; Fatigue; Ketamine
Keywords: Fatigue; Ketamine; Cancer
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Ketamine; Sodium Chloride; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Single intravenous dose given over 40 minutes
  Interventions: Drug: Ketamine; Drug: Placebo (saline)
- 2 (Active Comparator): Single intravenous dose goven over 40 minutes
  Interventions: Drug: Placebo (saline); Drug: Midazolam; Drug: Midazolam(placebo)

INTERVENTIONS:
Drug: Ketamine — Single intravenous dose
  Arms: 1
Drug: Placebo (saline) — Given intravenously over 40 minutes
Drug: Ketamine — Single intravenous dose given over 40 minutes
  Arms: 1
Drug: Midazolam — Given intravenously over 40 minutes
  Arms: 2
Drug: Midazolam(placebo) — Given intravenously over 40 minutes
  Arms: 2

SUMMARY:
Background:

- Fatigue is a common side effect of cancer and its treatment. No medications can treat this fatigue. Researchers want to see if the drug ketamine can improve fatigue after radiation therapy for cancer. They will compare the effects of ketamine on fatigue to midazolam, a sedative with similar effects.

Objectives:

- To better understand fatigue in people who completed radiation therapy for cancer. To look at the effects of a dose of ketamine on fatigue.

Eligibility:

- Adults 18 and older who completed radiation therapy for cancer and are enrolled in NIH protocol 08-NR-0132.

Design:

* Participants will be screened with medical history, physical exam, and blood and urine tests. They will complete questionnaires about their fatigue and take a breath alcohol test.
* The study is divided into 2 phases:
* During the first phase I visit, participants will have blood taken. They will talk about their fatigue and other symptoms. They will take thinking and handgrip strength tests. Then they will get either ketamine or placebo (midazolam) through an intravenous line, placed by a needle guided by a thin plastic tube into an arm vein.
* Participants will have a follow-up phone call within 1 day.
* Participants will have phase I visits 3, 7, and 14 days after infusion. For the 3- and 7-day visits, participants will take thinking and handgrip strength tests. They will complete questionnaires, talk about infusion side effects, and have blood taken. For the 14-day visit, they will talk about their fatigue and infusion side effects. They will start phase II that day.
* Phase II visits are the same as phase I, except that the 14-day visit is over the phone.

DETAILED DESCRIPTION:
Although the underlying mechanisms of fatigue have been studied in several disease conditions (Bower et al., 2002; Brola et al., 2007), the etiology, mechanisms, and risk factors remain elusive, and this symptom remains poorly managed. Fatigue is conceptualized as a multidimensional symptom which incorporates temporal, sensory, cognitive/mental, affective/emotional, behavioral, and physiological dimensions (Voss, et al., 2006). We recently observed increased levels of neutrophic factors (brain-derived neurotrophic factor (BDNF)), glial-cell line derived neurotrophic factor (GDNF) and synaptosomal-associated protein (SNAP) from the serum samples of fatigued prostate cancer men receiving external beam radiation therapy, suggesting that fatigue may be a component of depression and the N-methyl-D-aspartate (NMDA) receptors may be involved in fatigue intensification during cancer therapy. Ketamine is an NMDA receptor antagonist and has been reported to treat acute depression (Berman et al., 2000; Prommer, 2012; Aan Het Rot et al., 2012). Depression and cancer-related fatigue (CRF) are highly correlated during cancer therapy (Portenoy and Itri, 1999; Roscoe et al., 2002, Servaes et al., 2002, Aan Het Rot et al., 2012).

This double-blind, placebo-controlled, cross-over study will explore the effect of a single, intravenous dose of ketamine in providing immediate reduction of fatigue following radiation therapy. The primary objective of the study is to determine the immediate effect of a single intravenous dose of ketamine in reducing clinically-significant worsening of fatigue following radiation therapy. The secondary objectives of this study are to investigate the levels of cytokines (i.e., tumor necrosis factor-alpha (TNFalpha), insulin-like growth factor 1 (IGF-I), interleukin (IL)-6, IL-8, transforming growth factors (TGF)alpha and beta), neurotrophic factors (i.e., BDNF, GDNF, SNAP), metabolic (i.e., apoliprotein, arginine, arginase), and mitochondrial (i.e., oxygen consumption rate, glycolysis rate) markers from peripheral blood before and after treatment with ketamine or placebo and relate these levels to self-reported fatigue, depression, and health-related quality of life (HRQOL) scores. This study also aims to measure cognitive function and skeletal muscle strength of patients before and after treatment with ketamine or placebo and relate these findings with self-reported fatigue, depression, and HRQOL scores.

We will enroll 40 subjects who completed radiation therapy for cancer within at least 3 months. The primary outcome measure of the study is the change in self-reported fatigue score after receiving a single intravenous dose (0.5 mg/kg) of ketamine or placebo. The secondary outcomes of this study include: the cytokine profile (e.g. TNFalpha, IGF-I, IL-6, IL-8, TGFalpha and TGFbeta), neurotrophic factors (e.g. BDNF, GDNF), metabolic (i.e., apoliprotein, arginine, arginase), and mitochondrial markers (i.e., Complex I-V, manganese superoxide dismutase (MnSOD), oxygen consumption rate, glycolysis rate) from blood samples; cognitive function test scores; depression scores; HRQOL scores; and skeletal muscle strength of study participants before and after a dose of ketamine or placebo.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must be enrolled in 08-NR-0132.
* Had cancer as determined by diagnostic testing such as cytology and imaging and confirmed from the oncologist s progress notes or reference letter;
* At least 3 months following localized radiation therapy (e.g. intensity-modulated radiation therapy) for cancer;
* Total received radiation dose is 40-80 Gray (Gy);
* Able to provide written informed consent and must exhibit understanding of the study during the informed consent process by passing at least 80% of the consent quiz;
* Greater than or equal to18 years of age;
* FACT-F score should be <43, to reflect that the study subjects fatigue symptoms are worse than the general population (Cella et al., 2002).

In addition to the above inclusion criteria, in order to receive the study drug (ketamine or placebo), the subject must have the following during the randomization visit:

-No clinically significant abnormal laboratory tests (i.e. absolute neutrophil count <1.5 thousand (K) cells/(micro)L, platelet <75K cells/(micro)L, hemoglobin <9 grams per deciliter (g/dL).

EXCLUSION CRITERIA:

* Progressive or unstable disease other than cancer of any body system causing clinically significant fatigue (e.g. class IV congestive heart failure, end-stage renal disease, liver failure, stage IV chronic obstructive pulmonary disease) including patients with systemic infections (e.g., human immunodeficiency virus (HIV), active hepatitis); and those with chronic inflammatory disease (e.g. rheumatoid arthritis, systemic lupus erythematosus);
* Uncontrolled hypertension and those with left ventricular dysfunction;
* Current psychotic features or a diagnosis of Schizophrenia or any other psychotic disorder as defined in the Diagnostic and Statistical Manual (DSM-IV);
* Subjects with a history of DSM-IV drug or alcohol dependency or abuse (except for caffeine or nicotine dependence) within the preceding 3 months. In addition, subjects who currently are using illicit drugs (except for caffeine or nicotine) must not have used illicit substances in the 2 weeks prior to screen and must have a negative alcohol and drug (except for prescribed benzodiazepines) breathalyzer and urine test at screening, respectively;
* Subjects with clinical hypothyroidism or hyperthyroidism;
* Subjects with one or more seizures, hallucinations, disorientation without a clear and resolved etiology;
* Subjects with traumatic brain injury and/or post-traumatic stress disorder;
* Treatment with a reversible monoamine oxidase inhibitor (MAOI) within two weeks prior to study drug administration;
* Treatment with fluoxetine within five weeks or aripiprazole within three weeks before study drug administration;
* Treatment with any other concomitant medication known to interact with ketamine 14 days prior to study drug administration.
* Received total body irradiation or cranial irradiation for cancer;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12-13; Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Change in fatigue score | Pre-Post ketamine

SECONDARY OUTCOMES:
Cognition, muscle strength, depression | Pre-Post ketamine
Cytokines, neurotrophins, metabolic mark | Pre-Post ketamine

CONTACTS AND LOCATIONS:
Overall Officials: Leorey N Saligan, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States